CLINICAL TRIAL: NCT00559312
Title: A 6-week Randomized, Double-blind, Placebo-controlled, Crossover Study to Assess the Effect of Fluticasone 250μg/Salmeterol 50μg Combination (FSC 250/50) on Exertional Dyspnea in Patients With Symptomatic Mild COPD
Brief Title: The Effect of Fluticasone/Salmeterol Combination on Exertional Breathlessness in Patients With Mild COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCO110755
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: COPD
Keywords: mild COPD; dyspnea; exercise; combination therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FSC 250/50 (Experimental): fluticasone 250μg/salmeterol 50μg combination
  Interventions: Drug: fluticasone/salmeterol combination
- Placebo (Placebo Comparator): matched placebo inhaler
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fluticasone/salmeterol combination — Diskus inhaler, fluticasone 250μg/salmeterol 50μg, twice daily, 6-week duration
  Other Names: Advair 250/50
  Arms: FSC 250/50
Drug: placebo — Placebo Diskus inhaler, twice daily, 6-week duration
  Arms: Placebo

SUMMARY:
Even patients with milder COPD can have significant physiological abnormalities which become more pronounced during exercise, leading to intolerable breathing discomfort (dyspnea). While there is a compelling physiological rationale for the efficacy of inhaled corticosteroid/long-acting bronchodilator combination therapy [i.e., fluticasone 250μg/salmeterol 50μg (FSC250/50)] in moderate to severe COPD, little information is available on the potential impact of this therapy in milder symptomatic disease. This study will be the first to explore mechanisms of dyspnea and activity limitation in milder COPD and will determine if there is a sound physiological rationale for the use of FSC as therapy for this subpopulation.

ELIGIBILITY:
Inclusion Criteria:

* Stable mild COPD,
* FEV1/FVC<0.7 and FEV1>60% predicted,
* Activity-related dyspnea (i.e., Baseline Dyspnea Index focal score <9, MRC dyspnea scale >2),
* Cigarette smoking history ≥20 pack-years.

Exclusion Criteria:

* Presence of a significant disease other than COPD that could contribute to dyspnea and exercise limitation,
* Important contraindications to clinical exercise testing,
* Use of daytime oxygen,
* History of Asthma.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Dyspnea intensity (Borg rating at a standardized time during exercise) | 6 weeks

SECONDARY OUTCOMES:
Exercise endurance time | 6 weeks
Measurements of small airway function | 6 weeks
Exercise measurements of ventilation, breathing pattern, operating lung volumes and respiratory mechanics | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Respiratory Investigation Unit at Kingston General Hospital, Kingston, Ontario, Canada